CLINICAL TRIAL: NCT03972410
Title: Early Psychotherapeutic Intervention After Childbirth Trauma: Comparison Between EMDR and Supportive Expressive Dynamic Psychotherapy
Brief Title: Eye Movement Desensitization and Reprocessing vs Supportive Expressive Dynamic Psychotherapy for Childbirth Trauma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Turin, Italy (Other)
Collaborators: Ospedale San Paolo (Other); Humanitas Hospital, Italy (Other)
Responsible Party: Principal Investigator, luca ostacoli, Associate professor of clinical psychology, University of Turin, Italy
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EMDR 2018-04
Record Dates: First submitted 2019-05-30; First posted 2019-06-03 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Childbirth Problems; Post Traumatic Stress Disorder
Keywords: childbirth trauma; post-traumatic stress; depression; post-partum PTSD; EMDR; Supportive Expressive Dynamic Psychotherapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression | interventions — Eye Movement Desensitization Reprocessing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eye Movement Desensitization and Reprocessing (EMDR) (Experimental): The EMDR treatment will follow the EMDR Recent Birth Trauma Protocol. This protocol was recently developed by some of the colleagues collaborating in this research project (Catteneo et al., 2018). This EMDR protocol can be used to intervene immediately after birth, or at later times. The main purposes of early intervention is to prevent the onset and development of PTSD and Post-partum Depression in the mother during the months following childbirth and to facilitate mother-newborn bonding.
  Interventions: Behavioral: EMDR
- Supportive Expressive Dynamic Psychotherapy (SEDP) (Active Comparator): The SEDP treatment (Luborsky 1984; Book, 1998) is one of the most widespread treatments and can be considered the treatment as usual in Italian maternity wards. This intervention includes both supportive techniques (to create a positive, helpful and empathic relationship with the patient) and expressive techniques (aimed at helping the patient to express and to understand and change problems).
  Interventions: Behavioral: SEDP

INTERVENTIONS:
Behavioral: EMDR — 2-4 sessions individual 60-min-long treatment sessions of EMDR Recent birth trauma protocol
  Arms: Eye Movement Desensitization and Reprocessing (EMDR)
Behavioral: SEDP — 2-4 sessions individual 60-min-long treatment sessions of SEDP
  Arms: Supportive Expressive Dynamic Psychotherapy (SEDP)

SUMMARY:
There is increasing evidence that about 30% of women evaluate their childbirth as traumatic and that women could develop post-traumatic stress disorder (PTSD) in response to events of birth. The mean prevalence of post-partum PTSD (PP-PTSD) was reported as 3-4% in community samples and 15.7-18.95% in high-risk samples.

The primary aim is to investigate the effectiveness of Eye Movement Desesitization and Reprocessing (EMDR) in treating post-traumatic and postpartum depressive symptoms in women who had a traumatic childbirth as compared to Supportive Expressive Dynamic Psychotherapy (SEDP) as therapy as usual.

Secondary outcomes are:

* to evaluate the differences between EMDR and SEDP in preventing the onset of PTSD and Post-partum Depression after 3 months;
* to evaluate the effectiveness of EMDR and SEDP on anxiety and mother-child bonding; The subjects of the study will be 60 women who had a traumatic childbirth in the previous 2 days. Women with a Impact of Event Scale-Revised (IES-R) score > or = to 24 will be treated with 2-4 sessions of EMDR or with SEDP.

Two follow-up assessments will be scheduled: at 6-weeks post-partum (after the end of the psychotherapeutic intervention) and at 12-weeks post-partum.

DETAILED DESCRIPTION:
About 30% of women evaluate their childbirth as traumatic and 3-4% women could develop post-traumatic stress disorder (PTSD) in response to traumatic childbirth. There is also a high co-morbidity between post-traumatic stress symptoms and post-partum depressive symptoms.

The aims of the present research project are:

* to investigate the effectiveness of Eye Movement Desesitization and Reprocessing (EMDR) therapy in treating post-traumatic and post-partum depressive symptoms in women who have just experienced a traumatic childbirth as compared to Supportive Expressive Dynamic Psychotherapy (SEDP);
* to evaluate the differences between EMDR and SEDP in preventing the onset of PTSD and Post-partum Depression diagnoses after three-months post-partum;
* to evaluate the effectiveness of EMDR and SEDP on associated anxiety symptoms and on mother-child bonding both after the treatment and at the follow-up evaluation;
* to compare the effects of EMDR and SEDP on physiological indexes (i.e. HRV and skin conductance) measured during the first and last treatment sessions;
* to evaluate if these physiological indexes could predict the treatments outcome (e.g. respondents vs. non respondents).

The design of this study is a multicenter, randomized controlled clinical trial.

Patients will be consecutively recruited from three clinical centers:

* Sant'Anna Hospital, Città della Salute e della Scienza of Turin, Italy, affiliated with University of Turin, Italy.
* Humanitas San Pio X Hospital, Milan, Italy.
* San Paolo Teaching Hospital, Milan, Italy.

Participants The subjects of the study will be 60 women who have experienced a traumatic childbirth in the previous 2 days. Those who have a score on the Impact of the Event Scale - Revised (IES-R) equal or greater than 24 (in order to consider also sub threshold post-traumatic stress symptoms) will be asked for their participation in the study.

Assessments The psychological evaluation will be performed at baseline (T0), within the third day postdelivery, with a limited number of questionnaires, in order not to weigh down the patient given the context of urgency and hospitalization.

The following instruments will be administered:

* Impact of Event Scale-Revised (IES-R).
* The Edimburgh Post-natal Depression Scale (EPDS).
* Peritraumatic Dissociative Experiences Questionnaire (Marmar, 1996).

Two follow-up assessments will be scheduled in order to evaluate the outcomes of the psychotherapeutic interventions and to monitor symptoms levels over time:

* at 6-weeks post-partum (i.e. after the end of the psychotherapeutic intervention) (T1);
* at 12-weeks post- partum (T2).

During these follow-ups the following questionnaires will be administrated:

* Impact of Event Scale-Revised (IES-R);
* Edimburgh Post-natal Depression Scale (EPDS);
* Generalised Anxiety Disorder Assessment (GAD-7);
* Postpartum Bonding Questionnaire (PBQ);
* Mini-International Neuropsychiatric Interview-Plus (MINI-Plus; Sheehan et al., 1998).

Interventions All the participants, regardless of the type of treatment, will receive between 2 and 4 (according to women's availability) individual 60-min-long treatment sessions conducted over 4-5 weeks.

The first two sessions will be carried out before the woman's discharge from the maternity ward, and the next three sessions will be performed on an outpatient basis.

The EMDR treatment will follow the EMDR Recent Birth Trauma Protocol. This protocol can be used to intervene immediately after birth, or at later times. The main purposes of early intervention is to prevent the onset and development of PTSD and Postpartum Depression in the mother during the months following childbirth and to facilitate mother-newborn bonding.

The SEDP treatment is one of the most widespread treatments and can be considered the treatment as usual in Italian maternity wards. This intervention includes both supportive techniques (to create a positive, helpful and empathic relationship with the patient) and expressive techniques (aimed at helping the patient to express and to understand and change problems).

Physiological measures of psychotherapeutic process During the first and last treatment sessions, women will be asked to wear a simple wristband (similar to a wristwatch) that will monitor the physiological parameters of HRV and skin conductance for the entire duration of the session. These data will be then correlated with the outcome of the interventions detected at the follow-up assessments and with the clinical data obtained at the beginning and end of each session.

PRIMARY AND SECONDARY OUTCOMES The primary outcome of this study will be differences between EMDR and SEDP in reducing the IES- R and the EPDS clinical scores after treatment and at the 12-weeks post-partum follow-up.

Secondary outcomes of the studies are:

* to compare differences between EMDR and SEDP in preventing the onset of PTSD and Post-partum Depression diagnoses at the 12-weeks post-partum follow-up;
* to compare the effects of EMDR and SEDP on HRV and skin conductance measured during the first and last treatment sessions;
* to evaluate if these physiological indexes could predict the treatments outcome (e.g.respondents vs. non respondents).

ELIGIBILITY:
Inclusion Criteria:

* having experienced a traumatic childbirth (e.g. difficult delivery with obstetric and gynecological problems; woman's inability to tolerate the pain);
* a score on the lES-R > or = 24;
* good comprehension of spoken Italian;
* legal capacity to consent to the treatment;

Exclusion Criteria:

* having a baby hospitalized in Special Care Baby Unit or Neonatal Intensive Care Unit (NICU) or with a serious, unstable medical condition; (2) having experienced a stillbirth or a live birth;
* severe suicidality, including ideation, plan, and intent;
* current serious psychological and psychiatric disorders, including psychotic disorders,bipolar disorders, active substance abuse;
* presence of overt dementia;
* a serious, unstable medical condition.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-01-08 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Post-traumatic stress symptoms | 6 weeks post-partum
  Reduction of post-traumatic stress symptoms, as assessed by Impact of Event Scale -Revised (IES-R). Total score range 0-88. Cut-off for presence post-traumatic symptoms>=33.

SECONDARY OUTCOMES:
Post-partum depression symptoms | 6 weeks post-partum
  Reduction of post-partum depressive symptoms, as assessed by Edimburgh Post-natal Depression Scale (EPDS). Total score range: 0-30, cut-off score for possible depression =8.
  Possible Depression: 10 or greater
Post-traumatic stress disorder diagnosis | 12 weeks post-partum
  proportion of patients with a diagnosis of Post-traumatic stress disorder, as assessed with Mini-International Neuropsychiatric Interview-Plus.
Post-partum depression diagnosis | 12 weeks post-partum
  proportion of patients with a diagnosis of Post-partum depression, as assessed with Mini-International Neuropsychiatric Interview-Plus.

OTHER OUTCOMES:
mother-infant bonding | 6 weeks post-partum
  Levels of mother-infant bonding, as evaluated with Postpartum Bonding Questionnaire (PBQ)
mother-infant bonding | 12 weeks post-partum
  Levels of mother-infant bonding, as evaluated with Postpartum Bonding Questionnaire (PBQ). The PBQ has four subscales which reflect impaired bonding (Scale 1) (12 items, ranging from 0 to 60), rejection and anger (Scale 2) (7 items, scores ranging from 0 to 35), anxiety about care (Scale 3) (4 items,scores ranging from 0 to 20) and risk of abuse (Scale 4) (2 items,scores ranging from 0 to 10). Brockington et al. (2001) suggest cut-off scores to identify problematic bonding of 12 for Scale 1, 17 for Scale 2, 10 for Scale 3 and 3 for Scale 4.
anxiety symptoms | 6 weeks post-partum
  levels of anxiety symptoms, as evalueated with Generalized Anxiety Disorder Assessment (GAD-7). Total score ranges from 0 to 21. Scores of 5, 10, and 15 represent cut-points for mild, moderate, and severe anxiety, respectively.
anxiety symptoms | 12 weeks post-partum
  levels of anxiety symptoms, as evalueated with Generalized Anxiety Disorder Assessment (GAD-7). Total score ranges from 0 to 21. Scores of 5, 10, and 15 represent cut-points for mild, moderate, and severe anxiety, respectively.

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - Humanitas San Pio X Hospital, Milan
  - San Paolo Teaching Hospital, Milan
  - AOU Città della Salute e della Scienza di Torino - Sant'Anna Hospital, Torino

IPD SHARING:
Plan to Share IPD: No